CLINICAL TRIAL: NCT00257582
Title: Long-term Study of Cetirizine Dry Syrup in Children Suffering From Various Type of Cutaneous Disease Accompanied With Pruritus.
Brief Title: Study Of Cutaneous Disease Accompanied With Pruritus In Pediatrics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104915
Record Dates: First submitted 2005-11-21; First posted 2005-11-23 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-05

CONDITIONS: Pruritus
Keywords: cetirizine; various type of cutaneous disease accompanied with Pruritus; pediatrics
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Cetirizine Dry Syrup

SUMMARY:
To assess the safety of long-term use of cetirizine dry syrup in children with various type of cutaneous disease accompanied on pruritus.

ELIGIBILITY:
Inclusion Criteria:

* Chronic urticaria
* Eczema & dermatitis group
* Atopic dermatitis
* Prurigo group: Acute prurigo, Prurigo subacuta, Chronic prurigo
* Pruritus cutaneous: Systemic pruritus cutaneous, Topical pruritus cutaneous
* Giving informed consent
* Children who have 2 grades or more pruritus score when assessed by the investigator or sub-investigator with the criteria for the diurnal or nocturnal pruritus score in the patient diary.
* Children with a pruritus severity of "2.Mild" or severer on the first day of the treatment period.

Exclusion criteria:

* have a history of drug hypersensitivity
* are pregnant, lactating or possibly pregnant female children.
* have asthma that requires the treatment with corticosteroid.
* cannot avoid the use of external steroid classified into "strong", "strongest" or "very strong".
* have pruritus only on face and head.
* have inappropriate complication of dermal disorder that may influence on the evaluation of the study drug.
* are undergoing specific desensitization therapy or immunomodulation therapy or phototherapy.

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60
Dates: Start 2005-08

PRIMARY OUTCOMES:
To assess the safety

SECONDARY OUTCOMES:
-severity of pruritus -total pruritus score -daily main prurutus score -Severity of eruption -Patient global Improvement rating -Body temperature -Adverse events -Cetirizine serum concentrations

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site